CLINICAL TRIAL: NCT06078800
Title: Phase I Clinical Study on the Safety, Tolerance, Pharmacokinetics and Efficacy of Pan-KRAS Inhibitor YL-17231 in Patients With Advanced Solid Tumors With KRAS Mutation
Brief Title: A Study of YL-17231 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL-17231-002
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor
Keywords: Nonsmall-cell lung cancer（NSCLC）; Colorectal cancer（CRC）; Pancreatic carcinoma; KRAS mutation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YL-17231 (Experimental): YL-17231 will be administrated orally from 0.25mg QD, 0.5mg BID to 10mg BID in sequence during dose excalation part and selected doses in dose expansion part,for 21 consecutive days as a treatment cycle
  Interventions: Drug: YL-17231

INTERVENTIONS:
Drug: YL-17231 — After a screening period of approximately 14 days, eligible patients will receive oral YL-17231 once or twice daily until documented disease progression, unacceptable AEs, intercurrent illness preventing further administrations of study treatment, investigator's decision to withdrawal, the patient's consent of withdrawal, pregnancy, or for administrative reasons. Following the end of treatment, patients will continue to be followed for safety for 30 days. Patients who permanently discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient's consent of withdrawal, lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.
  Other Names: Pan-KRAS Inhibitor YL-17231

SUMMARY:
This is a phase 1 open label multicenter study to evaluate the maximum tolerance, safety, tolerance and PK of oral YL-17231 in patients with advanced solid tumors with KRAS mutation, so as to confirm the recommended phase 2 dose of YL-17231 and obtain the preliminary efficacy information of patients with advanced solid tumors with KRAS mutation.

DETAILED DESCRIPTION:
The study will be conducted in China to provide safety, efficacy and PK data. A dose escalation part 1 will be conducted to determine the MTD, DLTs, and part 2 will confirm the safety/tolerability of the recommended Phase 2 dose (RP2D), of YL-17231 given twice daily, in patients with advanced solid tumors to obtain preliminary efficacy information. PK samplings at single dose stage Day 1 and at steady-state conditions (Cycle 1, Day 14) will be performed.

ELIGIBILITY:
Inclusion Criteria:

The patients must meet all the following inclusion criteria to be eligible for enrollment in this trial:

1. Age between 18 and 75 years (inclusive), with no gender restriction.
2. Locally advanced or metastatic solid tumors diagnosed histologically and genomically confirmed with KRAS mutation, excluding patients with a clear KRAS wild-type test report in the case of pancreatic cancer.

   A. For patients with NSCLC, previous treatment failure based on platinum-based first-line therapy; B. For patients with colorectal cancer, previous experience with at least two lines of systemic therapy (patients with colorectal cancer and high microsatellite instability should have received PD-1 or PD-L1 therapy if clinically applicable); C. For patients with solid tumors other than NSCLC or colorectal cancer, at least one prior systemic treatment is required.
3. In the dose escalation phase, measurable or non-measurable tumor lesions are acceptable based on RECIST1.1 criteria; in the dose expansion phase, at least one measurable tumor lesion is required.
4. ECOG performance status (PS) of 0-1.
5. Estimated life expectancy of ≥3 months.
6. Good organ function levels:

   * Absolute neutrophil count (ANC) ≥1.5×109/L;
   * Platelet count (PLT) ≥100×109/L;
   * Hemoglobin (Hb) ≥90g/L (no blood transfusion within 14 days before screening);
   * Total bilirubin (TBIL) ≤1.5 times the upper limit of normal;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (≤5.0 times the upper limit of normal for patients with liver metastasis);
   * Serum creatinine (Cr) ≤1.5 times the upper limit of normal or creatinine clearance ≥50ml/min;
   * Left ventricular ejection fraction (LVEF) ≥50%;
   * Fridericia-corrected QT interval (QTcF) <450ms.
7. Washout period of ≥4 weeks for macromolecular agents and intravenous chemotherapy drugs, and ≥2 weeks for oral fluoropyrimidine and small molecule targeted drugs.
8. Fertile males and females must agree to use medically approved contraceptive measures during the study period and for 6 months following the last administration of the study drug.
9. Women of childbearing potential must have a negative pregnancy test within 7 days prior to the first administration of the study drug; patients must not be breastfeeding, and if the subject has already ceased breastfeeding at the time of study entry, breastfeeding must have been discontinued from the day of the first administration of the study drug till at least 30 days after last administration of the study drug .
10. No previous treatment with investigational drugs within 1 month prior to participation in this trial.
11. High compliance and willingness to complete the trial as assessed by the investigator, and ability to adhere to the study protocol.
12. Voluntary participation in this clinical trial, understanding of the study procedures, and ability to provide written informed consent.

Exclusion Criteria:

Patients with any of the following conditions are not eligible for enrollment in this study:

1. Uncontrollable third-space effusion (such as large amounts of pleural or ascitic fluid).
2. Grade 3 or 4 gastrointestinal bleeding or variceal bleeding requiring transfusion, endoscopy, or surgical intervention within the past 3 months.
3. Previous diagnosis of other malignancies within the past five years, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cured in situ cervical cancer.
4. Inability to swallow, chronic diarrhea, or intestinal obstruction that could affect medication intake and absorption.
5. History of significant neurological or psychiatric disorders.
6. Active hepatitis B (positive for hepatitis B surface antigen and/or hepatitis B core antibody with HBV-DNA ≥103 copies/mL or ≥200 IU/mL) or hepatitis C (positive for hepatitis C virus antibody and/or HCV-RNA).
7. History of immunodeficiency, including positive HIV test, acquired or congenital immunodeficiency disorders, organ transplantation, or allogeneic bone marrow transplantation.
8. Major surgical procedures (excluding biopsy) within the past 4 weeks prior to the first administration of the study drug, significant trauma, or the need for elective surgery during the study period, or radical radiotherapy within the past 4 weeks prior to the first administration of the study drug.
9. Moderate or severe cardiac diseases:

   * Myocardial infarction, angina, III/IV congestive heart failure, pericardial effusion, or uncontrolled severe hypertension (up to 150/90 mmHg or below) within the past 6 months prior to the first administration of the study drug;
   * Clinically significant electrocardiogram abnormalities, such as symptomatic or persistent atrial or ventricular arrhythmias, second or third-degree atrioventricular block, bundle branch block, or ventricular hypertrophy;
   * Significant abnormalities on echocardiography, such as moderate or severe valvular dysfunction, assessed based on institutional lower limits; patients with minimal or mild valve regurgitation (tricuspid, pulmonary, mitral, or aortic) can be included in this study;
   * Various factors that may increase the risk of QTcF prolongation or cardiac arrhythmia events, such as hypokalemia, congenital long QT syndrome, or concomitant use of drugs that may prolong the QT interval.
10. Untreated brain metastases that meet one or more of the following criteria:

    * Requiring corticosteroids or dehydration treatment (excluding the use of antiepileptic drugs after surgery or radiotherapy);
    * Presence of clinically significant symptoms;
    * Tumor stability after radiotherapy or surgery lasting no longer than 4 weeks. Asymptomatic or controlled stable patients with treated brain metastases are eligible for enrollment.
11. Unresolved treatment-related toxicity greater than Grade 1 according to CTCAE 5.0 at the start of study treatment (alopecia excluded).
12. Medical conditions that, in the opinion of the investigator, pose a serious risk to patient safety or could interfere with the patient's ability to complete the study, such as uncontrolled diabetes, thyroid disease, interstitial lung disease, severe active infections, or uncontrolled chronic infections, Child-Pugh Class B or C liver cirrhosis.
13. Other reasons deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DLTs | At the end of Cycle 1 (each cycle is 21 days)
  Dose limited toxicities
TEAEs | From day 1 after taking the investigational product till 30 days after withdrawal from the study
  Treatment emergent adverse events

SECONDARY OUTCOMES:
Cmax | From day 1 to the end of Cycle 2 (each cycle is 21 days)
  Peak plasma concentration
AUC | From day 1 to the end of Cycle 2 (each cycle is 21 days)
  Area under the plasma concentration versus time curve
Tmax | From day 1 to the end of Cycle 2 (each cycle is 21 days)
  Time to maximum plasma concentration
T1/2 | From day 1 to the end of Cycle 2 (each cycle is 21 days)
  Elimination half-life
The overall response rate (ORR) | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The overall response rate (ORR) will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1
DOR | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Duration of response
Disease control rate, DCR | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The percentage of cases with remission (PR+CR) and stable lesions (SD) after treatment
Progression free survival, PFS | From date of screening until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS, defined as the time from the first dose of study treatment to first documented progression
Overall survival, OS | From date of screening until the date of death from any cause, assessed up to 36 months
  The time from randomization to death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Xu Ruihua, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China